CLINICAL TRIAL: NCT02204384
Title: Plasma Glucose and Insulin Responses After Consumption of Breakfasts With Different Sources of Soluble Fiber in Type 2 Diabetes Patients: a Randomized Crossover Clinical Trial
Brief Title: Glycemic and Insulinemic Response With Different Sources of Soluble Fiber in Patients Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Mirela Jobim de Azevedo, PhD, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 140161
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Dietary Modification; Diabetes Mellitus Type 2; Insulin Tolerance; Diabetic Blood Glucose Monitoring
Keywords: Dietary fiber; Dietary Supplements; Type 2 diabetes; Postprandial Period; Plasma insulin; Plasma glucose; Area Under Curve; Soluble fiber
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HFD Meal: high fiber from food (Experimental): HFD Meal: high amount of fiber from diet food sources (total fiber 9.7g; soluble fiber 5.4g)
  Interventions: Other: HFD Meal: High fiber from food
- HFS Meal: High fiber from supplement (Experimental): HFS Meal: high amount of soluble fiber from guar gum supplement (HFS; total fiber 9.1g; soluble fiber 5.4g) - Fiber Mais, Nestlé
  Interventions: Dietary Supplement: HFS Meal: High fiber from supplement
- UF Meal: usual amount of fiber (Experimental): UF Meal: usual amount of fiber (total fiber 2.4g; soluble fiber 0.8g)
  Interventions: Other: UF Meal: usual amount of fiber

INTERVENTIONS:
Other: HFD Meal: High fiber from food — High amount of fiber from diet food sources (HFD; total fiber 9.7g; soluble fiber 5.4g)
  Other Names: HFD
  Arms: HFD Meal: high fiber from food
Dietary Supplement: HFS Meal: High fiber from supplement — High amount of soluble fiber from guar gum supplement (HFS; total fiber 9.1g; soluble fiber 5.4g) - sachet 5 g Fiber Mais, Nestlé Brasil, São Paulo, BR
  Other Names: HFS
  Arms: HFS Meal: High fiber from supplement
Other: UF Meal: usual amount of fiber — Usual amount of fiber (UF; total fiber 2.4g; soluble fiber 0.8g)
  Arms: UF Meal: usual amount of fiber

SUMMARY:
To compare the acute effect of soluble fiber intake from foods or supplement after a common meal on postprandial plasma glucose and insulin in patients with type 2 diabetes. The hypothesis is a meal with a high content of soluble fiber from food determines glycemic and insulinemic response similar to a meal with a high content of soluble fiber from supplement sources.

DETAILED DESCRIPTION:
Three breakfasts (high amount of fiber from diet food sources - HFD, high amount of soluble fiber from guar gum supplement - HFS and usual amount of fiber -UF), isocaloric and similar distribution of carbohydrates, proteins and lipids, the order of breakfasts randomly determined. Meals HFD and HFS have the same amount of fiber from different sources, origin in food and supplement respectively. Meal UF consist of the same foods meal HFS, but without the use of soluble fiber supplement and white bread instead of rye bread (low fiber content in relation to meals HFD and HFS). The supplement (Sachet 5g - Fiber Mais ®: 60% guar gum and 40% inulin) will be added to the plain water to meal HFD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes
* Body Mass Index (BMI) <= 35 kg / m²
* Hemoglobin A1c (HbA1c) <= 9%

Exclusion Criteria:

* Serum creatinine >2.0 mg/dL
* Digestive diseases (e.g. malabsorption)
* Severe autonomic neuropathy (presence of symptomatic postural hypotension, gastroparesis, diabetic diarrhea)
* Recent cardiovascular event
* Cachexia
* Psychiatric disorder with impairment of understanding
* Participating in other research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-08; Primary Completion 2016-03 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC 0-180min) for glycemic and insulinemic responses | Prior to the initial meal A, B and C and 30, 60,120,180 minutes postmeal

CONTACTS AND LOCATIONS:
Overall Officials: Mirela J Azevedo, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Carvalho CM, de Paula TP, Viana LV, Machado VM, de Almeida JC, Azevedo MJ. Plasma glucose and insulin responses after consumption of breakfasts with different sources of soluble fiber in type 2 diabetes patients: a randomized crossover clinical trial. Am J Clin Nutr. 2017 Nov;106(5):1238-1245. doi: 10.3945/ajcn.117.157263. Epub 2017 Aug 30. PMID 28855225